CLINICAL TRIAL: NCT05582278
Title: HAIC Combined With Lenvatinib and Tislelizumab Versus D-TACE Combined With Lenvatinib and Tislelizumab in Advanced Unresectable Hepatocellular Carcinoma
Brief Title: HAIC+Lenvatinib+Tislelizumab vs D-TACE+Lenvatinib+Tislelizumab for Unresectable HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wen Li (Other)
Responsible Party: Sponsor-Investigator, Wen Li, Attending physician, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11011
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Unresectable Hepatocellular Carcinoma
MeSH Terms: interventions — lenvatinib; tislelizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HAIC+lenvatinib+tislelizumab (Experimental): Hepatic Arterial Infusion Chemotherapy Combined With lenvatinib and tislelizumab
  Interventions: Drug: HAIC; Drug: Lenvatinib; Drug: tislelizumab
- D-TACE+lenvatinib+tislelizumab (Experimental): Transarterial chemoembolization with drug-eluting beads Combined With lenvatinib and tislelizumab
  Interventions: Drug: D-TACE; Drug: HAIC; Drug: Lenvatinib

INTERVENTIONS:
Drug: D-TACE — CalliSpheres (100-300 µm) loaded with pirarubicin for transarterial chemombolization: Typically, one vial of the beads was loaded with 60 mg pirarubicin. If blushed tumors is still visible after the embolization with one vial of beads, regular microspheres (8spheres) with diameters of 100-700 μm are additionally injected.
  Other Names: D-TACE+lenvatinib+tislelizumab
  Arms: D-TACE+lenvatinib+tislelizumab
Drug: HAIC — FOLFOX-based regimen for hepatic arterial infusion chemotherapy: oxaliplatin, 100 mg/m2 infusion for 2 hours; calcium levofolinate, 200 mg/m2 infusion for 1 hours; and 5-FU, 400 mg/m2 bolus infusion and then 2400 mg/m2 continuous infusion over 46 h.
  Other Names: HAIC+Lenvatinib+tislelizumab
Drug: Lenvatinib — 12 mg/d for bodyweight ⩾ 60 kg or 8 mg/d for bodyweight <60 kg
  Other Names: Targeted therapy
Drug: tislelizumab — tislelizumab 200 mg, every 3 weeks.
  Other Names: PD-1 inhibitors
  Arms: HAIC+lenvatinib+tislelizumab

SUMMARY:
Drug-eluting Bead-Transarterial chemoembolization (D-TACE) is the most widely used palliative treatment for hepatocellular carcinoma (HCC) patients. While a number of studies demonstrate poor effect of D-TACE for patients in Advanced Unresectable HCC. The investigators previous study also revealed similar results in Advanced Unresectable HCC patients treated with D-TACE. Recently, the investigators previous study demonstrated that, compared with D-TACE, hepatic arterial infusion chemotherapy (HAIC) may improve tumor response in Advanced Unresectable HCC. Thus, the investigators carried out this prospective nonrandomized control to demonstrate the superiority of HAIC-based combination therapy over D-TACE-based combination therapy.

DETAILED DESCRIPTION:
HCC is one of the most common malignant tumors with the worst prognosis. At present, except for liver transplantation, surgical resection is the most effective therapy for patients with HCC. However, many patients are found to have advanced cancer as soon as they were diagnosed and lose the opportunity of radical resection and treatments are limited.More and more clinical research failures have hit the investigators' hard, until a clinical study named IMbrave150, published in the New England Journal of Medicine in 2020. It has opened up a new era of combination therapy, breaking the pattern of only a single mode of advanced liver cancer for more than ten years, making the investigators realize that for the treatment of patients with advanced liver cancer, the single treatment effect is often very limited, and combination therapy is the future.The investigators recent research showed that HAIC Combined With Lenvatinib and Tislelizumab brings good results to patients with advanced HCC.To identify a more effective and safety way for treating potentially resectable HCC patients, this study is designed to compare the safety and efficacy between HAIC-based combination therapy and D-TACE-based combination therapy for those patients in Advanced Unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced unresectable hepatocellular carcinoma treated by D- TACE, or HAIC combined with Lenvatinib and Tislelizumab as initial treatment
* Age between 18 and 75 years
* Child-Pugh A or B liver function
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate hematologic blood counts (white blood cell count >3ⅹ109/L, absolute neutrophil count >1.5ⅹ109/L, platelet count >10ⅹ109/L, hemoglobin concentration >85 g/L
* No extrahepatic metastasis

Exclusion Criteria:

* Severe underlying cardiac, pulmonary, or renal diseases
* History of a second primary malignant tumor
* Incomplete medical data
* Loss to follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Tumor Response | 6-8 weeks
  The tumor responses were evaluated by measuring the longest diameter of target lesions according to response evaluation criteria in solid tumors.(RECIST) version 1.1
Overall survival | 24months
  Overall survival (OS) was measured from the initiation of transarterial therapy to the date of death or the last follow-up.
Progression-free survival | 24 months
  Progression-free survival (PFS) was measured from the initiation of transarterial therapy to the time of progression or recurrence or last follow-up
Cancer embolism withdraws | 6-8 weeks
  The degree of thrombosis withdrawal of the portal vein or hepatic vein(VP1-VP4 or I-IV).

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No